CLINICAL TRIAL: NCT04550117
Title: Intraspinal Pressure Monitoring for Acute Traumatic Spinal Cord Injury: A Validation Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre Foundation, Manitoba (Other)
Responsible Party: Principal Investigator, Perry Dhaliwal, Assistant Professor of Neurosurgery, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS23117 9B2019:075)
Record Dates: First submitted 2020-06-24; First posted 2020-09-16 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2023-12

CONDITIONS: Spinal Cord Injuries; Spine Injury
Keywords: spinal cord perfusion pressure; spinal cord injury; intraspinal pressure; spinal reactivity
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraspinal Pressure Monitoring (Experimental): A fiberoptic pressure monitoring device will be placed into the subarachnoid space at the site of traumatic spinal cord injury
  Interventions: Procedure: Insertion of Intraspinal pressure monitor

INTERVENTIONS:
Procedure: Insertion of Intraspinal pressure monitor — A fiberoptic pressure monitoring wire will be placed into the subarachnoid space at the site of traumatic spinal cord injury

SUMMARY:
Intraspinal pressure monitoring has been advanced as a potential technique for evaluating spinal cord perfusion after traumatic spinal cord injury. In this study, the investigators aim to validate the technique for insertion of a fiberoptic pressure monitoring device in the subarachnoid space at the site of injury for measurement of intraspinal pressure and spinal cord perfusion pressure. The primary objective of this study is to validate the methodology of invasive intraspinal pressure monitoring to derive parameters for optimal spinal cord perfusion pressure, spinal cord reserve capacity and spinal reactivity index using data obtained during the patient's stay in the intensive care unit.

Secondary objectives of this study will be to a) evaluate the safety of invasive intraspinal pressure monitoring, b) prospectively evaluate the overall relationship between spinal cord perfusion pressure and functional outcomes in patients with acute traumatic spinal cord injury and c) evaluate the relationship between spinal cord perfusion pressure, motor evoked potentials and functional outcomes after incomplete spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* • patients with acute traumatic spinal cord injury ASIA A, B or C

  * age between 18-70yrs

Exclusion Criteria:

* patients with central cord syndrome
* patients presenting to hospital >48hrs from time of spinal cord injury
* patients unable to communicate in english language
* pre-existing cognitive impairment
* penetrating spinal cord injury
* pre-existing neurodegenerative disorder involving brain or spinal cord
* patients with concomitant injuries requiring emergent surgical intervention

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Derivation of parameters for optimal spinal cord perfusion pressure using intraspinal pressure data | 1 year
  Derivation of parameters for optimal spinal cord perfusion pressure.

SECONDARY OUTCOMES:
Measurement of the accuracy of probe placement in relation to the site of injury | 1 year
Measure the correlation between spinal cord perfusion pressure and the American Spinal Injury Association (ASIA) Impairment scale, Quality of Life Index and Spinal Cord Independence Measure score. | 1 year
Record rates of adverse events in patients having insertion of intraspinal pressure monitor | 1 year
  Measure infection rates, rates of pseudomeningoceles, neurological injury, probe dislodgment, meningitis and or subdural hematoma at injury site.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dhaliwal P, Wilkinson M, Zeiler FA. The Winnipeg Intraspinal Pressure Monitoring Study (WISP): A protocol for validation of fiberoptic pressure monitoring for acute traumatic spinal cord injury. PLoS One. 2022 Sep 20;17(9):e0263499. doi: 10.1371/journal.pone.0263499. eCollection 2022. PMID 36126069